CLINICAL TRIAL: NCT01688531
Title: A Pilot Study to Investigate Filiation Between Primary and Secondary Lesions in Acne Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: RD.03.SPR.40183E; NCT01718665 (obsolete NCT alias)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2016-03

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD0271 0.1%/CD1579 2.5% gel (Experimental): Split-face design, one application a day for 6 months
  Interventions: Drug: CD0271 0.1%/CD1579 2.5% gel vehicle
- CD0271 0.1%/CD1579 2.5% gel vehicle (Placebo Comparator): Split-face design, one application a day for 6 months
  Interventions: Drug: CD0271 0.1%/CD1579 2.5% gel

INTERVENTIONS:
Drug: CD0271 0.1%/CD1579 2.5% gel — one application (pea-sized amount according to the labelling) on a half-face, 5 to 7 days for 6 months
  Arms: CD0271 0.1%/CD1579 2.5% gel vehicle
Drug: CD0271 0.1%/CD1579 2.5% gel vehicle — one application (pea-sized amount according to the labelling) on a half-face, 5 to 7 days for 6 months
  Arms: CD0271 0.1%/CD1579 2.5% gel

SUMMARY:
Exploratory, international, multi-centre, randomized, investigator blinded study in acne

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 35 years inclusive
* Subjects with active, moderate acne

Exclusion Criteria:

* The subject has a secondary acne form (chloracne, drug-induced acne, etc.) (Screening)
* The subject has a severity of acne that is not amenable to treatment with CD0271-CD1579 (Screening)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Description and documentation of acne lesions | over 6 months

SECONDARY OUTCOMES:
Treatment effect on acne lesions | over 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (2):
  - Galderma Investigational site, Windsor, Ontario
  - Galderma Investigational site, Montreal, Quebec
- Galderma Investigational site, Nantes, France